CLINICAL TRIAL: NCT04909502
Title: A Phase IIa, Open-label, Multicentre Dose-Finding Trial in Patients With Relapsing Forms of Multiple Sclerosis (RMS) to Evaluate the Safety, Tolerability and Preliminary Efficacy of EHP-101
Brief Title: Evaluation of Safety, Tolerability and Preliminary Efficacy of EHP-101 in Relapsing Forms of Multiple Sclerosis
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Temporary recruitment pause to re-assess the protocol design, specifically the eligibility criteria
Sponsor: Emerald Health Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EHP-101-MS02
Record Dates: First submitted 2021-05-14; First posted 2021-06-01 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-04

CONDITIONS: Relapsing Forms of Multiple Sclerosis
Keywords: Multiple Sclerosis; Nervous System Diseases; Demyelinating Autoimmune Diseases; Autoimmune Diseases of the Nervous System; Relapsing Forms of Multiple Sclerosis; Relapsing Remitting Multiple Sclerosis; Relapsing Secondary Progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Nervous System Diseases; Autoimmune Diseases of the Nervous System; Multiple Sclerosis, Relapsing-Remitting | interventions — BID protein, human

STUDY DESIGN:
Intervention Model Description: The study will initially be conducted with 2 treatment arms starting in parallel. Patients will initially receive a 25 mg OD or a 25 mg BID dose. After 28 days, each patient will increase to a 50 mg OD or 50mg BID dose level, respectively, if deemed to be safe by the investigator.
Masking Description: Open Label design
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- EHP-101 Once a day (OD) (Experimental)
  Interventions: Drug: EHP-101 25 mg OD; Drug: EHP-101 50 mg OD
- EHP-101 Twice a day (BID) (Experimental)
  Interventions: Drug: EHP-101 25 mg BID; Drug: EHP-101 50 mg BID

INTERVENTIONS:
Drug: EHP-101 25 mg OD — 25 mg OD during the first 28 Days of the trial
  Arms: EHP-101 Once a day (OD)
Drug: EHP-101 25 mg BID — 25 mg BID during the first 28 Days of the trial
  Arms: EHP-101 Twice a day (BID)
Drug: EHP-101 50 mg OD — After 28 Days of treatment with 25 mg OD, patients will escalate to 50 mg OD up to the end of the trial
  Arms: EHP-101 Once a day (OD)
Drug: EHP-101 50 mg BID — After 28 Days of treatment with 25 mg BID, patients will escalate to 50 mg BID up to the end of the trial
  Arms: EHP-101 Twice a day (BID)

SUMMARY:
The purpose of this trial is to evaluate the safety, tolerability, pharmacokinetics, and preliminary efficacy of EHP-101 in adult subjects with Relapsing Forms of Multiple Sclerosis (RMS).

DETAILED DESCRIPTION:
An interventional, open label, randomized design will be used to test safety, tolerability, pharmacokinetics, and preliminary efficacy of EHP-101 in 50 patients ≥ 18 and ≤ 55 years of age with documented RMS. There will be a screening period of up to 28 days, 168 days treatment period, and 28 days follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults aged 18 to 55 years at the time of consent;
* Confirmed diagnosis of MS according to the revised 2017 McDonald criteria;
* Relapsing forms of MS (RMS) including Relapsing-Remitting MS (RRMS) and active Secondary Progressive MS (SPMS);
* Patients must have experienced at least 1 of the following within 12 months prior to Visit 1: an acute clinical relapse, gadolinium-enhancing T1 lesions on brain or spinal cord magnetic resonance imaging (MRI), or new T2 lesion(s) on brain or spinal cord MRI;
* Neurologically stable with no evidence of clinical relapse of MS or corticosteroid treatment within 28 days prior to the first investigational product administration;
* Naïve to prior MS treatment or discontinuing current MS treatment due to (1) intolerability, (2) laboratory abnormalities, (3) current treatment perceived by the patient to be ineffective, (4) patient preference, or (5) based on investigator judgement to switch MS therapy;
* An EDSS score of 0 to 6.0 (inclusive) at screening and enrolment visit;
* Willing and able to provide informed consent and capable of understanding and complying with the protocol.

Exclusion Criteria:

* Primary progressive MS (PPMS) or non-active secondary progressive MS (SPMS);
* Relapse during the 28 days prior to first investigational product administration;
* Total lymphoid irradiation, T-cell or T-cell receptor vaccination, total body irradiation, or total lymphoid irradiation at any time;
* Treatment with alemtuzumab, mitoxantrone, cyclophosphamide or cladribine at any time;
* MS treatment that may impact the efficacy or safety assessment defined as follows:

  1. 52 weeks or less prior to first investigational product administration: Immunosuppressant agents (e.g., cyclosporine, methotrexate, mycophenolate)
  2. 36 weeks or less prior to first investigational product administration: CD20 depletion therapies such as rituximab, ocrelizumab, ofatumumab or others. Condition for inclusion of patients who had CD20 depletion therapies more than 36 weeks prior to the first investigational product administration: may only be included if there is no clinically relevant B cell depletion and possible safety risk to patients based on the Investigator's opinion.
  3. 12 weeks or less prior to first investigational product administration: natalizumab
  4. 8 weeks or less prior to first investigational product administration: dimethyl-fumarate fingolimod
  5. 4 weeks or less prior to first investigational product administration: corticosteroids intravenous immunoglobulin (IVIG) ozanimod, siponimod, or ponesimod glatiramer acetate interferons
  6. 2 weeks or less prior to first investigational product administration: teriflunomide. Subject must exhibit no active agent in serum levels; cholestyramine or activated charcoal washout may be used to achieve this;
* Any one of the following values for laboratory test at screening:

  1. Haemoglobin < 9 g/dL;
  2. Neutrophils < 1.0 x 10^9/L;
  3. Platelets < 75 x 10^9/L;
  4. Serum transaminases > 2.0 x upper limit of normal;
  5. Total bilirubin ≥ 1.5 x upper limit of normal;
  6. Thyroid-stimulating hormone level >10% above of the upper limit of normal;
  7. Estimated glomerular filtration rate ≤60 mL/min/1.73m2 (using the Cockcroft-Gault equation);
  8. Lymphocytes < 1 × 10^9/L;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-10-19 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of Treatment Emergent Adverse Events | 168 days (24 weeks)
  This safety outcome combines the measure of the number of subjects experiencing adverse events (AEs), the nature and severity of those AEs and their relationship to the study treatments

SECONDARY OUTCOMES:
Brain lesion activity measured by MRI | 168 days (24 weeks)
Disease progression measured by MS Functional Composite (MSFC) | 168 days (24 weeks)
  The MSFC consists of three assessments of walking speed, processing speed and finger dexterity. The scores are combined to provide a Z-score (number of standard deviations away from mean of a normal population) with lower scores representing greater abnormality
Disease progression measured by Expanded Disability Status Scale (EDSS) | 168 days (24 weeks)
  The EDSS is an ordinal scale used for assessing neurological impairment of MS based on a neurological examination. It consists of scores in each of seven functional systems (FS) and an ambulation score that are then combined to determine the EDSS [ranging from 0 (normal) to 10 (death due to MS)]. The FSs are the Visual, Brain Stem, Pyramidal, Cerebellar, Sensory, Bowel & Bladder, and Cerebral functions. The FSs and EDSS steps will be assessed in a standardized manner
Disease progression measured by Symbol Digit Modalities Test (SDMT) | 168 days (24 weeks)
  The SDMT measures the time to pair abstract symbols with specific numbers. The test requires elements of attention, visuoperceptual processing, working memory, and psychomotor speed. The score is the number of correctly coded items from 0-110 in 90 seconds. The total score provides a measure of the speed and accuracy of symbol-digit substitution
Disability status measured by MS Functional Composite (MSFC) | 168 days (24 weeks)
  The MSFC consists of three assessments of walking speed, processing speed and finger dexterity. The scores are combined to provide a Z-score (number of standard deviations away from mean of a normal population) with lower scores representing greater abnormality
Disability status measured by Expanded Disability Status Scale (EDSS) | 168 days (24 weeks)
  The EDSS is an ordinal scale used for assessing neurological impairment of MS based on a neurological examination. It consists of scores in each of seven functional systems (FS) and an ambulation score that are then combined to determine the EDSS [ranging from 0 (normal) to 10 (death due to MS)]. The FSs are the Visual, Brain Stem, Pyramidal, Cerebellar, Sensory, Bowel & Bladder, and Cerebral functions. The FSs and EDSS steps will be assessed in a standardized manner
Disability status measured by Symbol Digit Modalities Test (SDMT) | 168 days (24 weeks)
  The SDMT measures the time to pair abstract symbols with specific numbers. The test requires elements of attention, visuoperceptual processing, working memory, and psychomotor speed. The score is the number of correctly coded items from 0-110 in 90 seconds. The total score provides a measure of the speed and accuracy of symbol-digit substitution
Time to first relapse | 168 days (24 weeks)
Preliminary Annualized Relapse Rate (ARR) | 168 days (24 weeks)
Percent of patients who experience a relapse | 168 days (24 weeks)
Proportion of patients who remain qualified as relapse-free | 168 days (24 weeks)
Change in blood levels of neurofilament light chain (NfL) | Baseline, 28 Days, 56 Days, 84 Days, 112 Days, 140 Days, 168 Days

OTHER OUTCOMES:
Microstructural analysis and assessment of potential remyelination measured by Magnetization Transfer Ratio (MTR) | 168 days (24 weeks)
Assessment of white matter diffusivity and integrity measured by Diffusion Tensor Imaging (DTI) | 168 days (24 weeks)
VCE-004.8 plasma trough levels for all patients | 197 Days (28 weeks)
Pharmacokinetic profile of VCE-004.8 in terms of maximum observed plasma concentration (Cmax) | Day 1 (pre-dose) and at 0.5, 1, 2, 3, 4 and 6 hours post-dose on Day 1 and Day 28
Pharmacokinetic profile of VCE-004.8 in terms of area under the plasma concentration-time curve (AUC) | Day 1 (pre-dose) and at 0.5, 1, 2, 3, 4 and 6 hours post-dose on Day 1 and Day 28

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - North Central Neurology Associates, Cullman, Alabama
  - Fullerton Neurology and Headache Center, Fullerton, California
  - Accel Research Sites - Brain and Spine Institute of Port Orange, Port Orange, Florida
- St. Vincent's Hospital, Melbourne, Victoria, Australia